CLINICAL TRIAL: NCT00320255
Title: A Randomized, Double-blind, Placebo-controlled Study of Apixaban for the Prevention of Thromboembolic Events in Patients Undergoing Treatment for Advanced Cancer: A Phase 2 Pilot Study
Brief Title: A Phase 2 Pilot Study of Apixaban for the Prevention of Thromboembolic Events in Patients With Advanced (Metastatic) Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-027
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Thrombosis; Cancer; Pulmonary Embolism
Keywords: anticoagulant
MeSH Terms: conditions — Thrombosis; Neoplasms; Pulmonary Embolism | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1: Placebo (Placebo Comparator): Participants received placebo tablets once daily
  Interventions: Drug: Placebo
- Cohort 1: Apixaban, 5 mg (Placebo Comparator): Participants received apixaban as tablet, 5 mg, once daily
  Interventions: Drug: Apixaban
- Cohort 1: Apixaban, 10 mg (Active Comparator): Participants received apixaban as tablet, 10 mg, once daily
  Interventions: Drug: Apixaban
- Cohort 1: Apixaban, 20 mg (Active Comparator): Participants received apixaban as tablet, 20 mg, once daily
  Interventions: Drug: Apixaban
- Cohort 2: Placebo (Placebo Comparator): Participants in this cohort were admitted to the trial following the addition of a protocol amendment (Amendment 5), which removed the prohibition of inclusion of patients receiving chemotherapy with concomitant antiangiogenic therapy with bevacizumab. Patients received placebo once daily.
  Interventions: Drug: Placebo
- Cohort 2: Apixaban, 5 mg (Active Comparator): Participants in this cohort were admitted to the trial following the addition of a protocol amendment (Amendment 5), which removed the prohibition of inclusion of patients receiving chemotherapy with concomitant antiangiogenic therapy with bevacizumab. Patients received apixaban as tablet, 5 mg, once daily.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Oral tablets administered once daily in 5-, 10-, or 20-mg dose
  Other Names: BMS-562247
  Arms: Cohort 1: Apixaban, 10 mg; Cohort 1: Apixaban, 20 mg; Cohort 1: Apixaban, 5 mg; Cohort 2: Apixaban, 5 mg
Drug: Placebo — Oral tablets administered once daily
  Arms: Cohort 1: Placebo; Cohort 2: Placebo

SUMMARY:
The purpose of this study is to learn whether apixaban is well-tolerated and acceptable as anticoagulant therapy, when administered to patients with advanced or metastatic cancer and at increased risk for venous thromboembolic events. Demonstration of a favorable benefit:risk profile could lead to significant reduction in this serious and sometimes fatal complication of ongoing cancer and its treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Recipients of either first- or second-line chemotherapy for advanced or metastatic lung, breast, gastrointestinal, bladder, ovarian, or prostate cancer or myeloma, selected lymphomas, or cancer of unknown origin
* Able to begin study medication ≤6 weeks of starting either first- or second-line chemotherapy.
* Expected course of chemotherapy must have been ≥ 90 days after the start of chemotherapy
* Per Protocol Amendment 5, patients receiving bevacizumab were eligible to participate, provided that bevacizumab was used for indications approved by local country law

Key Exclusion Criteria:

* Women who are pregnant, breastfeeding
* History of deep vein thrombosis or pulmonary embolism
* Active bleeding or at high risk of bleeding
* Metastatic brain cancer
* Familial bleeding diathesis
* Serious hemorrhage requiring hospitalization, transfusion, or surgical intervention within 4 weeks of study entry
* Expected survival <6 months or an Eastern Cooperative Oncology Group performance status ≥3.
* Candidates for bone marrow transplantation within the 12-week treatment period or 30-day follow-up period
* Uncontrolled hypertension (systolic blood pressure >200 mm Hg and/or diastolic blood pressure >110 mm Hg
* Coagulopathy (international normalized ratio >1.5 or platelet count <100*10^9/L) if not yet receiving chemotherapy or <50*10^9/L if receiving chemotherapy). Platelet count must have been >100*10^9/L before starting study medication
* One or more of the following: alanine aminotransferase >3 times the upper limit of normal (ULN), total bilirubin >2*ULN, or calculated creatinine clearance <30 mL/min.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (8):
  - Arizona Cancer Center, Tucson, Arizona
  - Univ. Of Southern Calif. /Norris Comprehensive Cancer Center, Los Angeles, California
  - Dana-Farber Cancer Inst, Boston, Massachusetts
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School Of Medicine, New York, New York
  - University Of Rochester, Rochester, New York
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas
- Canada (4):
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec

REFERENCES:
- [Derived] Kahale LA, Matar CF, Tsolakian I, Hakoum MB, Barba M, Yosuico VE, Terrenato I, Sperati F, Schunemann H, Akl EA. Oral anticoagulation in people with cancer who have no therapeutic or prophylactic indication for anticoagulation. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD006466. doi: 10.1002/14651858.CD006466.pub7. PMID 34622445
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 130 participants were enrolled and randomized; however, 1 withdrew consent and 2 no longer met study criteria. Therefore, 127 participants were treated. Reasons Not Completed listed in the data table below were summarized for 127 participants who received treatment.
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Started | 30 | 32 | 30 | 33 | 2 | 3
Received Treatment | 29 | 32 | 29 | 32 | 2 | 3
Completed | 19 | 25 | 24 | 25 | 2 | 3
Not Completed | 11 | 7 | 6 | 8 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 4 | 0 | 0
Not completed — Poor compliance/noncompliance | 1 | 1 | 0 | 1 | 0 | 0
Not completed — No longer meets study criteria | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 3 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to receive treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg | Total
Number analyzed (Participants) | 30 | 32 | 30 | 33 | 2 | 3 | 130
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 17 | 28 | 19 | 17 | 1 | 3 | 85
  65 years and older but younger than 75 years | 8 | 4 | 9 | 8 | 1 | 0 | 30
  75 years and older | 5 | 0 | 2 | 8 | 0 | 0 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 17 | 13 | 0 | 2 | 64
  Male | 15 | 15 | 13 | 20 | 2 | 1 | 66
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 27 | 27 | 26 | 25 | 2 | 3 | 110
  Black/African American | 0 | 2 | 1 | 3 | 0 | 0 | 6
  Asian | 2 | 2 | 1 | 2 | 0 | 0 | 7
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 2 | 3 | 0 | 0 | 6

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Composite of Venous Thromboembolism (VTE) and All-cause Death
Description: VTE includes symptomatic deep vein thrombosis (DVT) and pulmonary embolism (PE). Any 1 of the following was considered diagnostic for DVT:
  * New or previously undocumented noncompressibility of 1 or more proximal venous segments of the legs on CUS
  * Constant intraluminal filling defects on 2 or more views on contrast venography in 1 or more venous segments in the legs or pelvis or involving the inferior vena cava.
  Any 1 of the following was considered diagnostic for PE:
  * Constant intraluminal filling defects in 2 or more views on pulmonary angiography
  * Sudden contrast cutoff of 1 or more vessels more than 2.5 mm in diameter on a pulmonary angiogram
  * A high probability VQ lung scan showing 1 or more segmental perfusion defects with corresponding normal ventilation (mismatch defect)
  * An abnormal VQ lung scan with satisfaction of either criterion 1 or 2
  * Abnormal spiral computed tomography scan showing thrombus in pulmonary vessels.
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 4 [3.9 to 31.7] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 1 [0.1 to 16.2] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

2. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis (DVT), Nonfatal Pulmonary Embolism (PE), and All-cause Death
Description: Any 1 of the following was considered diagnostic for DVT:
  * New or previously undocumented noncompressibility of 1 or more proximal venous segments (popliteal vein or higher) of the legs on CUS
  * Constant intraluminal filling defects on 2 or more views on contrast venography in 1 or more venous segments in the legs or pelvis or involving the inferior vena cava.
  Any 1 of the following was considered diagnostic for PE:
  * Constant intraluminal filling defects in 2 or more views on pulmonary angiography
  * Sudden contrast cutoff of 1 or more vessels more than 2.5 mm in diameter on a pulmonary angiogram
  * A high probability VQ lung scan showing 1 or more segmental perfusion defects with corresponding normal ventilation (mismatch defect)
  * An abnormal VQ lung scan (nonhigh probability) with satisfaction of either criterion 1 or 2
  * Abnormal spiral computed tomography scan showing thrombus in pulmonary vessels.
Time Frame: First dose to 30 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 3 [2.2 to 27.4] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

3. Secondary Outcome: Number of Participants With Composite of Venous Thromboembolism (VTE) and VTE-related Death
Description: as for outcome 1
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 4 [3.9 to 31.7] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 1 [0.1 to 16.2] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

4. Secondary Outcome: Number of Participants With Composite of Proximal Deep Vein Thrombosis (DVT), Nonfatal Pulmonary Embolism (PE), and Venous Thromboembolism (VTE)-Related Death
Description: VTE includes symptomatic DVT and PE. Any 1 of the following was considered diagnostic for DVT:
  * New or previously undocumented noncompressibility of 1 or more proximal venous segments of the legs on CUS
  * Constant intraluminal filling defects on 2 or more views on contrast venography in 1 or more venous segments in the legs or pelvis or involving the inferior vena cava.
  Any 1 of the following was considered diagnostic for PE:
  * Constant intraluminal filling defects in 2 or more views on pulmonary angiography
  * Sudden contrast cutoff of 1 or more vessels more than 2.5 mm in diameter on a pulmonary angiogram
  * A high probability VQ lung scan showing 1 or more segmental perfusion defects with corresponding normal ventilation (mismatch defect)
  * An abnormal VQ lung scan with satisfaction of either criterion 1 or 2
  * Abnormal spiral computed tomography scan showing thrombus in pulmonary vessels.
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 3 [2.2 to 27.4] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

5. Secondary Outcome: Number of Participants With All-Cause Death
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

6. Secondary Outcome: Number of Participants With Pulmonary Embolism (Fatal or Nonfatal)
Description: Any 1 of the following was considered diagnostic for PE:
  * Constant intraluminal filling defects in 2 or more views on pulmonary angiography
  * Sudden contrast cutoff of 1 or more vessels of greater than 2.5 mm in diameter on a pulmonary angiogram
  * A high probability VQ lung scan showing 1 or more segmental perfusion defects with corresponding normal ventilation (mismatch defect)
  * An abnormal VQ lung scan with satisfaction of either criterion 1 or 2
  * Abnormal spiral computed tomography scan showing thrombus in pulmonary vessels.
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Groups:
- Cohort 2: Apixiban, 5 mg: Participants in this cohort were admitted to the trial following the addition of a protocol amendment (Amendment 5), which removed the prohibition of inclusion of patients receiving chemotherapy with concomitant antiangiogenic therapy with bevacizumab. Patients received apixaban as tablet, 5 mg, once daily.
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixiban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 1 [0.1 to 17.8] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

7. Secondary Outcome: Number of Participants With Nonfatal Pulmonary Embolism
Description: Any 1 of the following was considered diagnostic for PE:
  * Constant intraluminal filling defects in 2 or more views on pulmonary angiography
  * Sudden contrast cutoff of 1 or more vessels more than 2.5 mm in diameter on a pulmonary angiogram
  * A high probability VQ lung scan showing 1 or more segmental perfusion defects with corresponding normal ventilation (mismatch defect)
  * An abnormal VQ lung scan with satisfaction of either criterion 1 or 2
  * Abnormal spiral computed tomography scan showing thrombus in pulmonary vessels.
Time Frame: First dose to 2 days following last dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 1 [0.1 to 17.8] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

8. Secondary Outcome: Number of Participants With Deep Vein Thrombosis
Description: Any 1 of the following was considered diagnostic for DVT:
  * New or previously undocumented noncompressibility of 1 or more proximal venous segments of the legs on CUS
  * Constant intraluminal filling defects on 2 or more views on contrast venography in 1 or more venous segments in the legs or pelvis or involving the inferior vena cava.
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 4 [3.9 to 31.7] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 1 [0.1 to 16.2] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

9. Secondary Outcome: Number of Participants With Distal Deep Vein Thrombosis
Description: as for outcome 8
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 1 [0.1 to 17.8] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

10. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis
Description: as for outcome 8
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 3 [2.2 to 27.4] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 0 [NA to NA] — No statistical analyses were conducted for Cohort 2.

11. Secondary Outcome: Number of Participants Who Died and With Adverse Events (AEs), Serious Adverse Events (SAEs), Bleeding AEs, and Discontinuations Due to AEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: First dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants
  Deaths | 2 | 1 | 0 | 0 | 0 | 0
  SAEs | 9 | 6 | 3 | 5 | 1 | 0
  Bleeding AEs | 6 | 15 | 11 | 12 | 1 | 2
  Discontinuations due to AEs | 7 | 4 | 4 | 4 | 1 | 0

12. Primary Outcome: Number of Participants With Composite of Confirmed Major Bleeding and Clinically Relevant Nonmajor (CRNM) Bleeding
Description: Major bleeding was defined as clinically overt bleeding accompanied by 1 or more of the following:
  * A decrease in hemoglobin of 20 g/L or more or
  * Required transfusion of 2 or more units of packed red blood cells or whole blood, or
  * Occurred in a critical site
  * Contributed to death.
  CRNM bleeding was defined as bleeding that did not meet the criteria for major bleeding but that, in routine clinical practice, would be considered relevant and not trivial by a patient and physician. Such bleeding satisfied a priori criteria defined by the ICAC, including:
  * Skin hematoma
  * Epistaxis that lasted for longer than 5 minutes, was repetitive, or led to an intervention
  * Hematuria that was macroscopic and either spontaneous or lasted for longer than 24 hours after instrumentation of the urogenital tract
  * Any other bleeding type that was considered to have clinical consequences.
Time Frame: From first dose to 2 days following last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort 2: Apixaban, 5 mg
Number analyzed (Participants) | 29 | 32 | 29 | 32 | 2 | 3
Participants | 1 [0.1 to 17.8] | 1 [0.1 to 16.2] | 1 [0.1 to 17.8] | 4 [3.5 to 29.0] | 2 [NA to NA] — No statistical analyses were conducted for Cohort 2. | 3 [NA to NA] — No statistical analyses were conducted for Cohort 2.

ADVERSE EVENTS:
Groups:
- Cohort : Apixaban, 5 mg: :Participants in this cohort were admitted to the trial following the addition of a protocol amendment (Amendment 5), which removed the prohibition of inclusion of patients receiving chemotherapy with concomitant antiangiogenic therapy with bevacizumab. Patients received apixaban as tablet, 5 mg, once daily.
Arm/Group | Cohort 1: Placebo | Cohort 1: Apixaban, 5 mg | Cohort 1: Apixaban, 10 mg | Cohort 1: Apixaban, 20 mg | Cohort 2: Placebo | Cohort : Apixaban, 5 mg
Serious Adverse Events (participants affected / at risk) | 9/29 | 6/32 | 3/29 | 5/32 | 1/2 | 0/3
Other Adverse Events (participants affected / at risk) | 24/29 | 28/32 | 24/29 | 30/32 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=29) | Cohort 1: Apixaban, 5 mg (N=32) | Cohort 1: Apixaban, 10 mg (N=29) | Cohort 1: Apixaban, 20 mg (N=32) | Cohort 2: Placebo (N=2) | Cohort : Apixaban, 5 mg (N=3)
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal tract hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 3 | 1 | 1 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal decompression (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=29) | Cohort 1: Apixaban, 5 mg (N=32) | Cohort 1: Apixaban, 10 mg (N=29) | Cohort 1: Apixaban, 20 mg (N=32) | Cohort 2: Placebo (N=2) | Cohort : Apixaban, 5 mg (N=3)
Anxiety (Psychiatric disorders) | 1 | 3 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 2 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 4 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 7 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 3 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 4 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 6 | 7 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 2 | 5 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 3 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 3 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 5 | 1 | 2 | 3 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 4 | 7 | 1 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 2 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 4 | 2 | 3 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 2 | 2 | 2 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 3 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Oedema peripheral (General disorders) | 3 | 2 | 2 | 2 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 2 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 1 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 3 | 2 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 2 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 1 | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 4 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 5 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 2 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 7 | 10 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 2 | 1 | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 2 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.